CLINICAL TRIAL: NCT03803254
Title: Hepatic Arterial Infusion Chemotherapy Plus Lenvatinib and Programmed Cell Death Protein-1 Antibody Versus Hepatic Arterial Infusion Chemotherapy Plus Lenvatinib for Advanced Hepatocellular Carcinoma
Brief Title: HAIC Plus Lenvatinib and PD-1 Antibody Versus HAIC Plus Lenvatinib for Advanced HCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government)
Responsible Party: Principal Investigator, Shi Ming, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCC-S058
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Lenvatinib; PD-1 Antibody; Oxaliplatin, 5-Fluorouracil and Leucovorin; Hepatic arterial infusion chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol; lenvatinib; spartalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC plus lenvatinib and PD-1 antibody (Experimental): Hepatic arterial infusion chemotherapy plus lenvatinib and programmed cell death protein-1 antibody
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Folfox Protocol; Drug: Lenvatinib; Drug: PD-1 antibody
- HAIC plus lenvatinib (Active Comparator): Hepatic arterial infusion chemotherapy plus lenvatinib
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Folfox Protocol; Drug: Lenvatinib

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
Drug: Folfox Protocol — Oxaliplatin , fluorouracil, and leucovorin
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
Drug: PD-1 antibody — 3mg/kg intravenously every 2 weeks
  Arms: HAIC plus lenvatinib and PD-1 antibody

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin plus lenvatinib and programmed cell death protein-1 antibody compared with lenvtinib Alone in patients with hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin plus lenvatinib for advanced hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
Hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin was effective and safe for hepatocellular carcinoma. Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma, and programmed cell death protein-1 (PD-1) antibody was effective and tolerable in patients with advanced hepatocellular carcinoma. No study has compared HAIC plus lenvatinib and PD-1 antibody with HAIC plus lenvatinib. Thus, the investigators carried out this prospective randomized control study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Eastern Cooperative Oncology Group performance status of 0 to 2
* with no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Objective Response Rate (ORR) | 12 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on mRECIST. CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference to the baseline sum of the diameters of target lesions.
Adverse Events | 12 months
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospita, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong